# Association between the Quantitative Assessment of Schistocytes in Peripheral Blood Smear and Prognosis of Patient Initially Diagnosed as HELLP Syndrome

#### **Thesis**

Submitted for partial fulfillment of Master Degree in

Obstetrics & Gynecology

### Presented by Shimaa Bakry Mohammed

M. B., B. Ch. 2009

Faculty of Medicine, Ain Shams University Work at Abu Sewair medical administration

## Under the supervision of Ass. Prof. Ahmed Hamdy Naguib

Assistant Professor of Obstetrics and Gynecology Faculty of Medicine, Ain Shams University

#### Lecturer. Ayman Abd El-Kader Mohamed

Lecturer of Obstetrics and Gynecology
Faculty of Medicine, Ain Shams University

#### Lecturer, Rasha Abd El-Rahman El-Gamal

Lecturer of Clinical and Chemical Pathology Faculty of Medicine, Ain Shams University

Faculty of Medicine
Ain Shams University
2016

Association between the Quantitative Assessment of Schistocytes in Peripheral Blood Smear and Prognosis of Patient Initially Diagnosed as HELLP Syndrome (Study results)

#### Results

The current study was conducted at Ain Shams University Maternity Hospital during the period between January2015 and December 2015. A total of 100 women with an initial diagnosis of HELLP syndrome were recruited in the study. Blood sample taken within 12hrs peripartum and patients followed up 48hrs after delivery and subdivided in to 2 groups according to improvement or deterioration after 48hrs after delivery. All results were collected, tabulated and statistically analyzed.

Table-4 and figures 8-10 show the initial characteristics of included women.

Table-4 Initial Characteristics of Included Women.

| Age (years) | |
|-------------------------|------------------|
| Range | 18 - 38 |
| $Mean \pm SD$ | $27.51 \pm 4.98$ |
| Parity | |
| Range | 0 - 5 |
| Median (IQR) | 1 (1 – 2) |
| Gestational Age (weeks) | |
| Range | 27 - 38 |
| $Mean \pm SD$ | $34.3 \pm 2.91$ |

SD standard deviation

IQR interquartile range [central 50% of ascendingly-ordered set of data]

Data presented as range, mean  $\pm$  SD; or range, median (IQR)

**Figure-8** Bar-Chart showing Maternal Age Distribution in Included Women .



**Figure-9** Pie-Chart showing Parity Distribution in Included Women .



**Figure-10** Bar-Chart showing Gestational Age Distribution in Included Women .



Table-5 and figures 11-18 show the initial clinical and laboratory data of included women.

**Table-5** Initial Clinical and Laboratory Data in Included Women .

| Initial Data | |
|---------------------------------|-----------------|
| Systolic Blood Pressure (mm Hg) | |
| Range | 170 - 240 |
| Median (IQR) | 180(170-190) |
| Diastolic Blood Pressure (mm | |
| Hg) | |
| Range | 90 - 150 |
| Median (IQR) | 100 (100 – 120) |
| Albuminuria | |
| 3+ | 41 (41%) |
| 4+ | 32 (32%) |
| 5+ | 27 (27%) |
| Hb Concentration (g/dl) | |
| Range | 6.5 - 9.8 |
| Median (IQR) | 8.7 (8 – 9) |
| Platelet Count (x 10,000 per | |
| mm <sup>3</sup> ) | |
| Range | 28 - 97 |
| Median (IQR) | 77 (67 – 85) |
| Serum ALT (u/l) | |
| Range | 91 - 895 |
| Median (IQR) | 200 (149 – 278) |
| Serum AST (u/l) | |
| Range | 79 – 779 |
| Median (IQR) | 179 (135 – 250) |
| Serum Total Bilirubin (mg/dl) | |
| Range | 1.2 - 7.9 |
| Median (IQR) | 2.3 (1.6 – 3.3) |
| Serum Creatinine (mg/dl) | |
| Range | 1.4 - 6.3 |
| Median (IQR) | 1.9 (1.8 – 2.1) |

IQR interquartile range [central 50% of ascendingly-ordered set of data] Data presented as range, median (IQR); or number (percentage) Hb hemoglobin

ALT alanine transaminase

AST aspartate transaminase

**Figure-11** Box-Plot Chart showing Initial Systolic and Diastolic Blood Pressure in Included Women .



**Figure-12** Pie-Chart showing Albuminuria in Included Women .



**Figure-13** Box-Plot Chart showing Initial Hb Concentration in Included Women .



**Figure-14** Box-Plot Chart showing Initial Platelet Count in Included Women .



Figure-15 Box-Plot Chart showing Initial Liver



Transaminases in Included Women.

**Figure-16** Box-Plot Chart showing Initial Serum Bilirubin and Creatinine in Included Women .



Table-6 and figures 17-21 show the clinical and laboratory data 48 hours postpartum in included women.

**Table-6** Clinical and Laboratory Data 48 hours Postpartum in Included Women .

| Data 48 hours Postpartum | |
|-------------------------------|-------------------|
| Systolic Blood Pressure (mm | |
| Hg) | 110 - 230 |
| Range | 135 (120 – 185) |
| Median (IQR) | |
| Diastolic Blood Pressure (mm | |
| Hg) | |
| Range | 60 - 130 |
| Median (IQR) | 90 (70 – 100) |
| Hb Concentration (g/dl) | |
| Range | 5 – 13.3 |
| Median (IQR) | 9.7 (7.12 – 11) |
| Platelet Count (x 10,000 per | |
| mm <sup>3</sup> ) | |
| Range | 20 - 303 |
| Median (IQR) | 115 (65 – 135) |
| Serum ALT (u/l) | |
| Range | 7 – 2165 |
| Median (IQR) | 55 (25 – 281.5) |
| Serum AST (u/l) | |
| Range | 7 – 2143 |
| Median (IQR) | 36 (15 – 250) |
| Serum Total Bilirubin (mg/dl) | |
| Range | 0.1 - 10 |
| Median (IQR) | 1.3 (1.1 – 1.8) |
| Serum Creatinine (mg/dl) | |
| Range | 0.5 - 14.5 |
| Median (IQR) | 0.75 (0.6 - 2.75) |

IQR interquartile range [central 50% of ascendingly-ordered set of data]

Data presented as range, median (IQR)

Hb hemoglobin

ALT alanine transaminase

AST aspartate transaminase

Figure-17 Box-Plot Chart showing Systolic and Diastolic





Blood Pressure 48 hours Postpartum in Included Women. **Figure-18** Box-Plot Chart showing Hb Concentration 48 hours Postpartum in Included Women.

Figure-19 Box-Plot Chart showing Platelet Count 48 hours



Postpartum in Included Women .

**Figure-20** Box-Plot Chart showing Liver Transaminases 48 hours Postpartum in Included Women .



Figure-21 Box-Plot Chart showing Serum Bilirubin and



Creatinine 48 hours Postpartum in Included Women. Of the included 100 women, 25 (25%) women showed clinical and laboratory deterioration 48 hours postpartum. All women who deteriorated postpartum received plasma exchange. Of the included 100 women, 3 (3%) died (table-7, figures 22-23).

**Table-7** Postpartum Deterioration and Mortality in Included Women .

| Postpartum Deterioration | |
|---------------------------------------|----------|
| Yes | 25 (25%) |
| No | 75 (75%) |
| Received Plasma Exchange-<br>steroids | |
| Yes | 25 (25%) |
| No | 75 (75%) |
| Maternal Mortality | |
| Yes | 3 (3%) |

No 97 (100%)

Data presented as number (percentage)

Figure-22 Pie-Chart showing Postpartum Deterioration in Included Women.



**Figure-23** Pie-Chart showing Maternal Mortality in Included Wome .



There were no significant differences between women who deteriorated postpartum and women who did not regarding age, parity or gestational age (table-8, figures 24-26).

**Table-8** Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial Characteristics.

| | | Women who<br>Deteriorated | Women who Did not Deteriorate | P |
|---|---|---|---|---|
| | | Postpartum | Postpartum | |
| | | (n=25) | (n=75) | |
| Age (years) | | | | |
| Range | | 18 - 35 | 18 - 38 | 0.621* |
| $Mean \pm SD$ | | $27.08 \pm 4.58$ | $27.65 \pm 5.13$ | NS |
| Parity | | | | |
| Range | | 1 - 4 | 0 - 5 | 0.972** |
| Median (IQR) | | 1(1-2) | 1 (1 – 2) | NS |
| Gestational | Age | | | |
| (weeks) | - | | | |
| Range | | 27 - 38 | 27 - 38 | 0.407* |
| $Mean \pm SD$ | | $33.88 \pm 3.14$ | $34.44 \pm 2.83$ | NS |

SD standard deviation

IQR interquartile range [central 50% of ascendingly-ordered set of data]

Data presented as range, mean  $\pm$  SD; or range, median (IQR)

- \* Analysis using Independent Student's t-test
- \*\* Analysis using Mann-Whitney's U-Test NS non-significant

Figure-24 Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Maternal Age.

**Figure-25** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did not regarding Parity.



**Figure-26** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Gestational Age .

There were no significant differences between women who deteriorated postpartum and women who did not regarding the initial values of systolic blood pressure, diastolic blood pressure, albuminuria, hemoglobin concentration, platelet count or serum creatinine. The initial levels of serum ALT, AST and total bilirubin were, however, significantly, higher in women who deteriorated postpartum (table-9, figures 27-34).

**Table-9** Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial Clinical and Laboratory Data.

| Initial Data | Women who Deteriorated Postpartum (n=25) | Women who Did not<br>Deteriorate Postpartum<br>(n=75) | P |
|---|---|---|---|
| Systolic Blood Pressure (mm Hg) | | | |
| Range | 170 – 190 | 170 - 240 | 0.366* |

#### Association between the Quantitative Assessment of Schistocytes in Peripheral Blood Smear and Prognosis of Patient Initially Diagnosed as HELLP Syndrome (Study results)

| Median (IQR) | 180 (170 – 190) | 180 (170 – 190) | NS |
|---|---|---|---|
| Diastolic Blood Pressure (mm Hg) | | | |
| Range | 100 - 130 | 90 – 150 | 0.123* |
| Median (IQR) | 100(100-110) | 110(100-120) | NS |
| Albuminuria | | | |
| 3+ | 13 (52%) | 28 (37.7%) | |
| 4+ | 5 (20%) | 27 (36%) | 0.287** |
| 5+ | 7 (28%) | 20 (26.7%) | NS |
| Hb Concentration (g/dl) | | | |
| Range | 6.6 - 9.5 | 6.5 - 9.8 | 0.747* |
| Median (IQR) | 8.6(7.5 - 9.05) | 8.7 (8 – 9) | NS |
| Platelet Count (x 10,000 per mm <sup>3</sup> ) | | | |
| Range | 41 - 90 | 28 – 97 | 0.285* |
| Median (IQR) | 70 (58 – 85) | 78 (67 – 85) | NS |
| Serum ALT (u/l) | | | |
| Range | 91 – 895 | 95 – 494 | 0.043* |
| Median (IQR) | 287 (145 – 448) | 196 (155 – 233) | S |
| Serum AST (u/l) | | | |
| Range | 87 – 779 | 79 – 515 | 0.004* |
| Median (IQR) | 256 (155 – 430) | 170 (125 – 224) | S |
| Serum Total Bilirubin (mg/dl) | | | |
| Range | 1.4 - 7.9 | 1.2 - 5.2 | <0.001* |
| Median (IQR) | 3.4(2.4-4.2) | 1.9(1.6-2.7) | HS |
| Serum Creatinine (mg/dl) | | | |
| Range | 1.5 - 6.3 | 1.4 - 3.8 | 0.105* |
| Median (IQR) | 2(1.8-2.3) | 1.9 (1.8 – 2) | NS |

IQR interquartile range [central 50% of ascendingly-ordered set of data]
Data presented as range, median (IQR); or number (percentage)
\* Analysis using Mann-Whitney's U-Test

NS non-significant – S significant – HS highly significant

<sup>\*\*</sup> Analysis using Chi-squared Test

Figure-27 Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Initial Systolic Blood Pressure.

Figure-28 Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Initial Diastolic Blood Pressure.

**Figure-29** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial Hemoglobin Concentration.



**Figure-30** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial Platelet Count .



Figure-31 Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Initial ALT.

**Figure-32** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial AST .



**Figure-33** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did not regarding Initial Serum Total Bilirubin .



Figure-34 Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Initial Serum Creatinine .

The median schistocytes percentage was significantly higher in women who showed postpartum deterioration, when compared to women who did not deteriorate (table-10, figure-35).

**Table-10** Difference between Women who Deteriorated Postpartum and Women who did not regarding Schistocytes Percentage .

| | Women who<br>Deteriorated<br>Postpartum<br>(n=25) | Women who Did<br>not Deteriorate<br>Postpartum<br>(n=75) | P |
|---|---|---|---|
| Schistocytes (%) | | | |
| Range | 0 - 44 | 0 - 6 | <0.001* |
| Median (IQR) | 5.5(2-8.4) | 0.5(0.05-0.7) | HS |

IQR interquartile range [central 50% of ascendingly-ordered set of data] Data presented as range, median (IQR)

<sup>\*</sup> Analysis using Mann-Whitney's U-Test HS highly significant

**Figure-35** Box-Plot Chart showing Difference between Women who Deteriorated Postpartum and Women who did



not regarding Schistocytes Percentage.

The median schistocytes percentage was significantly higher in women who died when compared to women who survived (table-11, figure-36).

**Table-11** Difference between Women who Died and Women who Survived regarding Schistocytes Percentage.

| | Women who Died (n=3) | Women who Survived (n=97) | P |
|---|---|---|---|
| Schistocytes (%) | | | |
| Range | 8.3 - 44 | 0 - 39 | <0.001* |
| Median (IQR) | 39(8.3-44) | 0.5(0.1-1.1) | HS |

IQR interquartile range [central 50% of ascendingly-ordered set of data]

Data presented as range, median (IQR)

\* Analysis using Mann-Whitney's U-Test

HS highly significant

**Figure-36** Box-Plot Chart showing Difference between Women who Died and Women who Survived regarding Schistocytes Percentage .



Receiver operator characteristic (ROC) curve was constructed for schistocytes percentage as a predictor of postpartum deterioration in included women. The curve showed a significant predictability as denoted by the significantly large area under the curve (AUC) (figure-37).

**Figure-37** ROC Curve for Schistocytes Percentage as Predictor of Postpartum Deterioration in Included Women .



AUC = 0.883, 95% CI (0.770 to 0.996), p<0.001

Table-15 shows the validity of schistocytes at different cutoff values as predictor of postpartum deterioration.

**Table-12** Validity of Schistocytes as Predictor of Postpartum Deterioration in Included Women.

| Schistocy | Sensitivi | Specifi | PPV | NPV | FP | FN | LR+ |
|-----------|-----------|---------|------|------|------|----|-----|
| tes | ty | city | | | | | |
| | | | 66.7 | 95.5 | 14.7 | 12 | 6 |
| ≥ 0.95% | 88% | 85.3% | % | % | % | % | |
| | | | 87.5 | 94.7 | 4% | 16 | 21 |
| ≥ 1.4% | 84% | 96% | % | % | | % | |
| | | | 95.2 | 93.7 | 1.3% | 20 | 60 |
| ≥1.9% | 80% | 98.7% | % | % | | % | |

PPV positive predictive value -NPV negative predictive value FP false positive -FN false negative-LR+ positive likelihood ratio

ROC curves were constructed for initial clinical and laboratory data as predictors of postpartum deterioration. Among all measured variables, only initial ALT, initial AST and initial total bilirubin were significant predictors of postpartum deterioration. Their AUCs, though being significantly large, were smaller than the AUC for

schistocytes; indicating that the latter is a more significant and better predictor for postpartum deterioration (figure-38). **Figure-38** ROC Curves for Initial Clinical and Laboratory Data as Predictors of Postpartum Deterioration in Included Women.



Initial SBP: AUC = 0.441, 95% CI (0.324 to 0.559), p=0.381 Initial DBP: AUC = 0.404, 95% CI (0.283 to 0.525), p=0.152 Initial Hb Concentration: AUC = 0.479, 95% CI (0.341 to 0.616), p=0.750

Initial Platelet Count: AUC = 0.429, 95% CI (0.293 to 0.564), p=0.286

Initial ALT: AUC = 0.636, 95% CI (0.484 to 0.787), p=0.043 Initial AST: AUC = 0.694, 95% CI (0.553 to 0.834), p=0.004 Initial Serum Total Bilirubin: AUC = 0.772, 95% CI (0.656 to 0.887), p=0.001

Initial Serum Creatinine: AUC = 0.607, 95% CI (0.468 to 0.746), p=0.110

Table-13 shows the validity of initial values of ALT, AST, and total bilirubin as predictors of postpartum deterioration. Again, the validity parameters were remarkably lower than the corresponding parameters of schistocytes.

**Table-13** The validity of initial values of ALT, AST, and total bilirubin as predictors of postpartum deterioration.

| | Sensitivity | Specificit | PPV | NPV | FP | FN | LR |
|---|---|---|---|---|---|---|---|
| | | y | | | | | + |
| Initial ALT | | | | | | | |
| $\geq$ 230 u/L | 60% | 72% | 41.7 | 84.4 | 28% | 40% | 2.1 |
| | | | % | % | | | |
| Initial AST | | | | | | | |
| $\geq$ 240 u/L | 60% | 84% | 55.6 | 86.3 | 16% | 40% | 3.8 |
| | | | % | % | | | |
| <b>Initial Total</b> | | | | | | | |
| Bilirubin≥ | 68% | 81.3% | 54.8 | 88.4 | 18.7 | 32% | 3.6 |
| 2.95 mg/dl | | | % | % | % | | |

ALT alanine transaminase - AST aspartate transaminase

PPV positive predictive value -NPV negative predictive value

FP false positive -FN false negative

LR+ positive likelihood ratio

ROC curve was constructed for schistocytes percentage as a predictor of maternal mortality in included women. The curve showed a significant predictability as denoted by the significantly large area under the curve (AUC) (figure-39).

**Figure-39** ROC Curve for Schistocytes Percentage as Predictor of Maternal Mortality in Included Women .



AUC = 0.985, 95% CI (0.956 to 1.103), p=0.004

Table-14 shows the validity of schistocytes as predictor of maternal mortality in included women.

**Table-14** Validity of Schistocytes as Predictor of Maternal Mortality in Included Women .

| Schistoc vtes | Sensiti<br>vity | Specifi<br>city | PP<br>V | NP<br>V | FP | F<br>N | LR<br>+ |
|---|---|---|---|---|---|---|---|
| ≥ 8.2% | 100% | 95.9% | 42.9 | 100 | 4.1 | 0 | 24. |
| | | | % | % | % | % | 3 |

PPV positive predictive value NPV negative predictive value FP false positive FN false negative LR+ positive likelihood ratio

There were significant positive correlations between schistocytes percentage and each of systolic and diastolic blood pressures, serum ALT, serum AST, serum total bilirubin and serum creatinine 48 hours postpartum. There were significant negative correlations between schistocytes and each of hemoglobin concentration and platelet count 48 hours postpartum (table-15, figures 40-43).

**Table-15** Correlation between Schistocytes and Both Clinical and Laboratory Data 48 hours Postpartum in Included Women .

| Data 48 hours Postpartum | Sch | Schistocytes |
|--------------------------|-------|--------------|
| Systolic Blood Pressure | $r_s$ | 0.479 |
| | P | < 0.001 |
| | | HS |
| | | 0.439 |
| Diastolic Blood Pressure | $r_s$ | < 0.001 |
| | P | HS |
| Hb Concentration | $r_s$ | -0.527 |
| | P | < 0.001 |
| | | HS |
| Platelet Count | $r_s$ | -0.406 |
| | P | < 0.001 |
| | | HS |

| Serum ALT | rs | 0.373 |
|-----------------------|-------|---------|
| | P | < 0.001 |
| | | HS |
| Serum AST | $r_s$ | 0.353 |
| | P | < 0.001 |
| | | HS |
| Serum Total Bilirubin | $r_s$ | 0.313 |
| | P | 0.002 |
| | | S |
| Serum Creatinine | rs | 0.411 |
| | P | < 0.001 |
| | | HS |

Hb hemoglobin ,ALT alanine transaminase

AST aspartate transaminase

r<sub>s</sub> Spearman's rank correlation coefficient

HS highly significant - S significant

**Figure-40** Scatter-Plot Chart showing Correlation between Schistocytes and Platelet Count 48 hours Postpartum in Included Women.



**Figure-41** Scatter-Plot Chart showing Correlation between Schistocytes and ALT 48 hours Postpartum in Included Women .



**Figure-42** Scatter-Plot Chart showing Correlation between Schistocytes and Total Bilirubin 48 hours Postpartum in Included Women .



**Figure-43** Scatter-Plot Chart showing Correlation between Schistocytes and Serum Creatinine 48 hours Postpartum in Included Women .



 $Association\ between\ the\ Quantitative\ Assessment\ of\ Schistocytes\ in\ Peripheral\ Blood\ Smear\ and\ Prognosis\ of\ Patient\ Initially\ Diagnosed\ as\ HELLP\ Syndrome\ (Study\ results)$